CLINICAL TRIAL: NCT06911957
Title: The Impact of Chronic Consumption of Plant-based Fibres on Cognitive Performance, Gut Microbiome and Mental Health Outcomes in Older Adults: a Pilot Randomised Controlled Trial
Brief Title: PRECOG Pilot Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Collaborators: Biotechnology and Biological Sciences Research Council (Other); Myota Limited (Unknown); i-NutriLife Hub (Unknown)
Responsible Party: Principal Investigator, Piril Hepsomali, Principle Investigator, University of Reading
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: UREC 25/03
Record Dates: First submitted 2025-03-20; First posted 2025-04-04 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Cognition; Affect (Mental Function); Gut Microbiome
Keywords: prebiotics; cognition; depression; anxiety; gut microbiome diversity; relative abundance
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active: prebiotic blend (powder) (Experimental): Subjects will consume 10g of prebiotic fibre powder in their tea/coffee/water at breakfast.
  Interventions: Dietary Supplement: Prebiotic blend
- Active: matched placebo (powder) (Placebo Comparator): Subjects will consume 10g of matched placebo powder in their tea/coffee/water at breakfast.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Prebiotic blend — 10g of prebiotic fibre blend powder
  Arms: Active: prebiotic blend (powder)
Dietary Supplement: Placebo — 10g of matched placebo powder
  Arms: Active: matched placebo (powder)

SUMMARY:
This pilot study aims to investigate the chronic effects of a prebiotic blend on cognitive, affective and gut microbiome outcomes in healthy adults aged 60-75 years.

DETAILED DESCRIPTION:
This pilot study will employ a double-blind, randomised, placebo-controlled parallel design to investigate the chronic effects of 12-week-long prebiotic blend consumption on cognitive, affective, gut microbiome, metabolic, and anthropometric outcomes in healthy older adults with mild to moderate subjective cognitive complaints. Fifty participants will be randomised to Intervention or Placebo groups where they will be consuming 10g of prebiotic fibre blend or 10g of placebo (matched placebo powder) per day for 12-weeks. Outcome measures will be acquired before and after a 12-week chronic supplementation. These will include cognitive measures of overall cognitive functioning, and domain-specific cognitive performance, affective measures of depression and anxiety symptomatology; gastrointestinal symptomatology; systolic and diastolic blood pressure, as well as height, weight, hip and waist circumference. In addition, stool samples will be collected at all timepoints to assess microbiome diversity and composition.

ELIGIBILITY:
Inclusion Criteria:

* Aging between 60-75 years old
* Having normal vision and hearing
* Having a normal body mass index (BMI<30)

Exclusion Criteria:

* Having mild to moderate subjective cognitive complaints
* Smoking
* Having food allergies
* Following restrictive and/or unbalanced diets
* Changing dietary intake majorly in past month
* Being diagnosed with any psychiatric or neurologic conditions (e.g. schizophrenia, depression, dementia) including eating disorders
* Being diagnosed with any cardiometabolic diseases (including type II diabetes and cardiovascular disease), or suffering from hypertension or thrombosis related disorders or suffer from thyroid disease
* Currently taking anticoagulants, antiplatelet medication, antidepressants, proton-pump inhibitors
* Currently consuming prebiotic or probiotic supplements
* Continuous antibiotic use for > 3 days within 1 month prior to enrolment
* Continuous use of weight-loss drug for > 1 month before screening
* Having a significant gastrointestinal (GI) condition affecting absorption including (but not limited to) inflammatory bowel disease; total colectomy or bariatric surgery; irritable bowel disease; end stage renal disease; active cancer, or treatment for any cancer, in last 3 years
* Having a high fibre intake defined as > 20g of fibre/day
* Wheat and/or gluten intolerance and having coeliac disease

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Cognitive Drug Research Computerized Assessment System (COGDRAS) scores | From baseline (pre intervention) to week 12 (post intervention)
  The COGDRAS battery consists of 8 individual cognitive tests testing memory, attention and reaction times.
Gut microbiome diversity | From baseline (pre intervention) to week 12 (post intervention)
  Stool samples will be collected to measure gut microbiome diversity. Indices of alpha and beta diversity will be analysed (16s sequencing).
Gut microbiome composition | From baseline (pre intervention) to week 12 (post intervention)
  Stool samples will be collected to measure gut microbiome composition (genus and species) (16s sequencing).

SECONDARY OUTCOMES:
Geriatric Depression Scale scores | From baseline (pre intervention) to week 12 (post intervention)
  A validated self-report measure of depression that includes 15-items.
Geriatric Anxiety Inventory scores | From baseline (pre intervention) to week 12 (post intervention)
  A validated self-report measure of anxiety that includes 20-items.
Montreal Cognitive Assessment (MoCA) score | From baseline (pre intervention) to week 12 (post intervention)
  Composite measure of global cognitive function
Gastrointestinal Symptom Rating Scale Scores | From baseline (pre intervention) to week 12 (post intervention)
  A validated self-report measure of gastrointestinal symptoms that includes 15-items (combined into five symptom clusters depicting Reflux, Abdominal pain, Indigestion, Diarrhoea and Constipation) .
Blood Pressure | From baseline (pre intervention) to week 12 (post intervention)
  Systolic and diastolic blood pressure (in mmHg) will be measured.
Positive and Negative Affect Schedule (PANAS) | From baseline (pre intervention) to week 12 (post intervention)
  A 20-item questionnaire measuring positive and negative affect.
Hip and waist circumference | From baseline (pre intervention) to week 12 (post intervention)
  Hip and waist circumference (in cm) will be measured.
Body Mass Index | From baseline (pre intervention) to week 12 (post intervention)
  Weight (in kg) and height (in m) will be combined to report BMI in kg/m^2.

OTHER OUTCOMES:
Telephone Interview for Cognitive Status-40 | Baseline (pre intervention)
  A questionnaire that assesses cognitive status. It will be used to screen participants. Only individuals who score between 6 and 20 (depicting mild to moderate subjective cognitive complaints) will be included in the study.
FiberScreen Scores | Baseline (pre intervention)
  A questionnaire that assesses fibre intake. It will be used to screen participants. Individuals who adhere to a high fibre diet (>20g fibre/day) will be excluded from the study.
EPIC Norfolk Food Frequency Questionnaire (FFQ) | Baseline (pre intervention)
  The FFQ is a validated tool for gauging the average habitual dietary intake of micro and macronutrients of an individual in the UK. Data will be processed using the FETA software.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Reading, School of Psychology and Clinical Languages, Reading, Berkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No